CLINICAL TRIAL: NCT03823586
Title: AQUApay (AQUA Predictive Ability in Youths): Study on the Predictive Ability of the Questionnaire AQUA© in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, Coordinator of the group "Clinical and Environmental Epidemiology of Pulmonary and Allergic Pediatric Diseases". Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: 01/2019
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Young Athletes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children
  Interventions: Diagnostic Test: Questionnaire AQUA©, pediatric version
- Adolescents
  Interventions: Diagnostic Test: Questionnaire AQUA©, pediatric version

INTERVENTIONS:
Diagnostic Test: Questionnaire AQUA©, pediatric version — A version of AQUA© recently adapted and pretested in young athletes. It is a self-administered questionnaire composed of 25 items includes items about type, duration and intensity of training sessions, allergic status, habits of children (supplements and drugs intake) and their parents (smoking), presence and burden of infections.

SUMMARY:
Allergic diseases like asthma, rhinitis, conjunctivitis and dermatitis are very frequent in athletes, even if those complaining allergic symptoms do not always receive a medical diagnosis. Many athletes already start competitive sport activities in pediatric age, but allergy screening tests are usually not performed when assessing eligibility to sport practice. Therefore, the objective of the present study is assessing the predictive ability of the Allergy Questionnaire for Athletes (AQUA©), pediatric version, to predict the atopic status in young athletes.

ELIGIBILITY:
Inclusion Criteria:

- Athletes, males or females, 7 to 14 years old

Exclusion Criteria:

* Use of systemic antihistamines or long term or high dose corticosteroids in the last two weeks;
* Poor understanding of written or spoken Italian;
* Lack of written informed consent.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Athletes aged 7 to 14 years old, recruited from several sport associations located in the city of Palermo (Italy).
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Atopic status | Day 0
  Having at least 1 positive skin prick test to common aero-allergens

SECONDARY OUTCOMES:
Psychological well-being | Day 0
  Percentage score from the WHO-5 questionnaire for measuring psychological well-being.
  The questionnaire is composed of 5 questions scored on a scale ranging from 0 (worse outcome) to 5 (best outcome). The total (raw) score is obtaining by summing all the individual score items, therefore it ranges from 0 (worse outcome) to 25 (best outcome). To obtain a percentage score ranging from 0 to 100, the raw score is multiplied by 4. A percentage score of 0 represents worst possible outcome, whereas a score of 100 represents best possible outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology (IBIM), National Research Council, Palermo, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fasola S, Ferrante G, Malizia V, Bommarito N, Del Giacco S, Bonini M, Baiardini I, Bellafiore M, La Grutta S. Validity and repeatability of the Pediatric Allergy Questionnaire for Athletes (AQUAped) for the screening of atopy. Pediatr Allergy Immunol. 2021 Apr;32(3):437-444. doi: 10.1111/pai.13410. Epub 2020 Dec 2. PMID 33202069